CLINICAL TRIAL: NCT01687790
Title: The Assessment of Molecular Breast Imaging (MBI) in Distinguishing Benign From Malignant Breast Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Christiane Hakim, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO12030005
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-07

CONDITIONS: Breast Abnormalities
Keywords: molecular breast imaging; breast disease; breast biopsy
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- molecular breast imaging (Experimental)
  Interventions: Device: molecular breast imaging (Discovery)

INTERVENTIONS:
Device: molecular breast imaging (Discovery)
  Other Names: Discovery NM750b

SUMMARY:
The primary hypothesis of this project is that using molecular breast imaging (MBI) in evaluating women with equivocal mammographic or sonographic findings will demonstrate high specificity in distinguishing benign from malignant breast disease and, as a result, decrease the number of biopsies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Women who have indeterminate mammographic or sonographic findings who are recommended and for biopsy

Exclusion Criteria:

* Known contraindication to mammographic imaging
* women who are pregnant
* women who are lactating
* women who have significant existing breast trauma
* women who have breast implants
* Women under 18 years of age.
* women who had previous benign breast surgery within 1 year
* Males and children
* Women who are unable to understand or execute written informed consent
* Women who refuse to have a biopsy
* Women with any known renal disease - if an MRI is deemed necessary, a serum creatine will be checked prior to injection of contrast. Using the National Kidney Foundation recommendations, a glomerular filtration rate (GFR) greater than 60 may safely receive intravenous gadolinium-based MRI contrast. Those individuals with a GFR >30 and <60 can receive the contrast but at a reduced dose (typically half). Those with a GFR <30 will not receive MRI contrast and will not undergo the exam. Breast MRI must be done with contrast if evaluating for cancer. Several factors can affect the GFR such as age, body size, creatinine, renal status and will be calculated from the blood drawn. GFR is the final determinant and a creatinine greater than 1.6 usually has a GFR that precludes a Breast MRI with contrast. The final determinant will be the GFR.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Hakim, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: single group
Groups:
- Molecular Breast Imaging: molecular breast imaging (Discovery)
Period: Overall Study
Arm/Group | Molecular Breast Imaging
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Women scheduled for biopsy based on a suspicious mammogram and/or ultrasound. MBI results were compared to pathology.
Arm/Group | Molecular Breast Imaging
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 13
Age, Continuous [Median (Full Range); unit: years] | 56 [33 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Specificity of MBI. Specificity is Defined as the Number of True Negatives/ Total Number of Negative Pathology Results.
Description: The number of indeterminate lesions with negative MBI uptake and negative/benign pathology results.Reported are number of indeterminate lesions with negative MBI uptake and negative/benign pathology results (true negatives).
Time Frame: 1 year
Population: Analysis population included the number of indeterminate lesions that had negative/benign pathology results.
Measure: Number; unit: lesions
Groups:
- Molecular Breast Imaging: Participants received molecular breast imaging before biopsy
Arm/Group | Molecular Breast Imaging
Number analyzed (Participants) | 42
lesions | 27

2. Secondary Outcome: Sensitivity of MBI. Sensitivity in This Case is Defined as the Number of True Positives/ Total Number of Positive Pathology Results.
Description: Reported are the number of indeterminate lesions with marked, moderate, or mild uptake and positive pathology results (true positives).
Time Frame: 1 year
Population: Analysis population included the number of indeterminate lesions that had positive pathology results.
Measure: Number; unit: lesions
Arm/Group | Molecular Breast Imaging
Number analyzed (Participants) | 20
lesions | 19

ADVERSE EVENTS:
Arm/Group | Molecular Breast Imaging
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No